CLINICAL TRIAL: NCT01066312
Title: Investigating the Accuracy of Manual Muscle Testing for Distinguishing Congruent From Incongruent Statements Under Varying Levels of Blinding
Brief Title: The Accuracy of Manual Muscle Testing
Status: Completed | Type: Observational
Sponsor: Parker Research Institute (Other)
Responsible Party: Principal Investigator, Dr. Anne M. Jensen, DPhil Candidate, Parker Research Institute
Other Study IDs: MMT Study
Record Dates: First submitted 2010-02-09; First posted 2010-02-10 (Estimated); Last update posted 2017-06-19 (Actual); Status verified 2017-06

CONDITIONS: Lying
Keywords: Muscle testing; Kinesiology; Muscles; Complementary and Alternative Medicine; Practitioner Experience; This study is actually not a randomised controlled trial,; but an assessment of diagnostic test accuracy. We will be; looking at the accuracy of MMT to distinguish congruent from; incongruent statements under varying levels of blinding.
MeSH Terms: conditions — Deception

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Practitioners: Healthcare practitioners who either use, have used or do not use MMT in practice
- Testees: Healthy adults with no experience with MMT

SUMMARY:
Manual Muscle Testing (MMT) practiced by over a million practitioners worldwide. However, it's accuracy under varying levels of blindness has not yet been considered. This study will test this accuracy.

Study Hypothesis: MMT can accurately distinguish congruent from incongruent statements. Also, the accuracy of MMT is positively correlated with practitioner experience.

DETAILED DESCRIPTION:
Manual Muscle Testing is a non-invasive assessment tool used by millions of healthcare practitioners worldwide for a variety of purposes. First described in the literature by Lovett and Wight in 1915, MMT was originally used to assess muscular weakness in polio victims. In 1949, physiotherapists Kendall and Kendall refined MMT into an art and science with the publication of their benchmark text, Muscles: Testing and Function. This type of MMT is still used today to assess neuromuscular integrity.

In the 1960's, a different use for MMT was described by Dr. George Goodheart. In Goodheart's technique, called Applied Kinesiology (AK), MMT is used to evaluate a variety of additional functions of the body, apart from neuromuscular integrity. From Goodheart's work, many different techniques have emerged which use this second type of MMT. Moreover, it is estimated that over one million healthcare practitioners worldwide use this type of MMT: medical doctors, dentists, chiropractors, osteopaths, physiotherapists, other health professionals - plus even some lay-persons.

As a result of this divergence, there exists two very different forms of MMT: (1) orthopaedic muscle testing to quantify muscle strength and asses neurological integrity, and (2) the other type of muscle testing - which called be called "muscle response testing" which is used to obtain additional information about a patient. What that information is depends upon the MMT system being used and what information is sought. It is this latter form of MMT that this proposed study will investigate. Therefore, for the remainder of this application, the term "MMT" will be used to refer only to the second type ("muscle response testing").

The basic premise of MMT is that when there is some aberrant nervous system input to a muscle, it is less likely to be able to resist an external force. During a manual muscle test, an external force is applied to one muscle or group of muscles which at first causes an isometric then an eccentric contraction. Consequently, the muscle being tested is labelled "weak" or "strong" based on its ability to resist this external force.

A number of different techniques use MMT to test the body's physiological response to semantic stimuli, which may have both cognitive and emotional components. Monti et al. found that a MMT following congruent statements yielded significantly different results compared to a MMT following incongruent statements. A congruent statement is one that the person believes is true. An incongruent statement is one the person believes is false. The study by Monti et al. used self-referential statements similar to this study design, however they used statements such as, "My name is (insert one's name)". One criticism of using this type of self-referential statements is that in all likelihood both the muscle tester and the muscle testee know the verity of the statement, therefore, they are both unblinded, which may have introduced biased. While it is generally accepted by those who use this assessment tool that some bias exists in MMT, little is currently known about the degree of this bias. Therefore the main objective of this study is to investigate the accuracy of MMT to distinguish congruent from incongruent statements under varying degrees of blindness.

A further aim of this study are to explore if practitioner experience correlate with MMT accuracy. Caruso and Leisman reported greater MMT accuracy in experienced practitioners compared to inexperienced practitioners. Therefore, this study will test the reproducibility of these findings.

There will be two groups of participants selected for this study: (1) Practitioners, and (2) Testees - where the Practitioner will perform MMT on the Testee as the Testee speaks a statement. The Testee will know if s/he is speaking a true or false statement. However, for some statements, the Practitioner will be blind to the verity of the statement.

Results will be analysed for percent correct - that is, percent of muscle tests which accurately predicted the verity of the spoken statement.

ELIGIBILITY:
Inclusion Criteria:

1. Practitioners

   * health care provider
   * aged between 18 and 65 years old
   * healthy
   * fluent in English
2. Testees

   * aged between 18 and 65 years old
   * healthy
   * fluent in English

Exclusion Criteria:

1. Practitioners

   * a current physical disability or injury of either upper extremity
   * Blind, deaf or mute
2. Testees

   * a current physical disability or injury of either upper extremity
   * Prior experience with MMT
   * Blind, deaf or mute
   * are known to the Practitioner

NOTE: For this study, no compensation is possible.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Practitioenrs - Healthcare providers - healthy adults
  2. Testees - Healthy adults with no prior experience with MMT
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2010-03 (Actual); Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Percent correct | 1 hour

SECONDARY OUTCOMES:
Practitioner Experience | 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Anne M Jensen, DC, MS, MSc, Principal Investigator — Parker Research Institute
Locations (1):
- Parker Research Institute, Dallas, Texas, United States

REFERENCES:
- [Background] Caruso W, Leisman G. A force/displacement analysis of muscle testing. Percept Mot Skills. 2000 Oct;91(2):683-92. doi: 10.2466/pms.2000.91.2.683. PMID 11065332
- [Background] Caruso W, Leisman G. The clinical utility of force/displacement analysis of muscle testing in applied kinesiology. Int J Neurosci. 2001;106(3-4):147-57. doi: 10.3109/00207450109149745. PMID 11264916
- [Background] Ludtke R, Kunz B, Seeber N, Ring J. Test-retest-reliability and validity of the Kinesiology muscle test. Complement Ther Med. 2001 Sep;9(3):141-5. doi: 10.1054/ctim.2001.0455. PMID 11926427
- [Background] Pollard H, Lakay B, Tucker F, Watson B, Bablis P. Interexaminer reliability of the deltoid and psoas muscle test. J Manipulative Physiol Ther. 2005 Jan;28(1):52-6. doi: 10.1016/j.jmpt.2004.12.008. PMID 15726035
- [Background] Bossuyt PM, Reitsma JB, Bruns DE, Gatsonis CA, Glasziou PP, Irwig LM, Lijmer JG, Moher D, Rennie D, de Vet HC; STARD Group. Towards complete and accurate reporting of studies of diagnostic accuracy: the STARD initiative. Fam Pract. 2004 Feb;21(1):4-10. doi: 10.1093/fampra/cmh103. PMID 14760036
- [Derived] Jensen AM, Stevens RJ, Burls AJ. Estimating the accuracy of muscle response testing: two randomised-order blinded studies. BMC Complement Altern Med. 2016 Nov 30;16(1):492. doi: 10.1186/s12906-016-1416-2. PMID 27903263